CLINICAL TRIAL: NCT02862379
Title: Evaluation of a Personalized Rehabilitation Program for Elderly Patients That Fall : Impact on the Fear of Falling
Brief Title: Personalized Rehabilitation Program for Elderly Patients That Fall
Acronym: CHUTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC-P0034
Record Dates: First submitted 2016-08-01; First posted 2016-08-11 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Elderly; Falls; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elderly patients that fall (Experimental): Personalized rehabilitation program for elderly patients that fall for the first time. This intervention is a home-based program combining exercises, home modifications and education on fall risk factors.
  Interventions: Behavioral: home-based program

INTERVENTIONS:
Behavioral: home-based program — The objective of the rehabilitation program is to reduce the risk of falls after management of the risk factors identified. This intervention is a home-based program combining exercises, home modifications and education on fall risk factors

SUMMARY:
The risk of falling affects more than one third of people over 65 years old and over 50% of persons over 80 years. These falls have important consequences for the autonomy of the elderly patient and also increase the risk of sequelae and death.

The goal of this study is to evaluate a personalized rehabilitation program for elderly patients that fall for the first time and to measure the impact on the fear of falling of these patients. This intervention is a home-based program combining exercises, home modifications and education on fall risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Persons who have fallen minimum twice the last year
* 60 years old or more
* Mini Mental State Examination (MMSE) equal or superior to 23/30
* Persons who gave consent to participate in the study
* Persons with severe visual or hearing impairment

Exclusion Criteria:

* Patients with severe disease that might interfere with walking or with program monitoring

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Falls Efficacy Scale (FES-I) | Change from baseline at 6 months and 12 months
  The FES is a 10-item validated questionnaire that can be self-administered or completed during an interview. The person is asked to indicate on a 10-level rating scale his/her level of confidence in his/her capacity to accomplish a variety of activities of daily life (e.g., going up and down the stairs, taking a bath or shower) without falling. A FES score is calculated by adding up the score of each item.

SECONDARY OUTCOMES:
Number of falls the previous year before inclusion | at baseline
Life Space Assessment scale | Change from baseline at 6 months and 12 months
Get up and go test | Change from baseline at 6 months and 12 months
  It uses the time that a person takes to rise from a chair, walk three metres, turn around, walk back to the chair, and sit down. During the test, the person is expected to wear their regular footwear and use any mobility aids that they would normally require
Walking and talking test | Change from baseline at 6 months and 12 months
Tinetti test | Change from baseline at 6 months and 12 months
  It is a clinical test for assessing a person's static and dynamic balance abilities
Measure of the time that the patient is able to stay in station bipedal standing feet together followed by a monopodal support | Change from baseline at 6 months and 12 months
EuroQol five dimensions questionnaire (EQ-5D) | Change from baseline at 6 months and 12 months
  Questionnaire about quality of life
Incidence of falls during one year | through the study completion, an average of 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Romagny, Principal Investigator — ESPRAD CHUTE, GHICL
Locations (1):
- Esprad Chute, Ghicl, Lomme, France

IPD SHARING:
Plan to Share IPD: No